CLINICAL TRIAL: NCT07235761
Title: The Effect of Simulation Based Nursing Interventions on Mothers Prevention and Intervention of Home Accidents: A Randomized Controlled Trial
Brief Title: Preventing Home Accidents With Simulation Based Training
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Merve Şen, Specialist nurse, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SELCUKUNI-NURSING-2024-86
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Accident at Home; First Aid Training; Simulation Training
Keywords: Accident at home; First aid training; Simulation

STUDY DESIGN:
Intervention Model Description: This study employs a parallel group pretest posttest randomized controlled experimental design.
Who Masked: Outcomes Assessor
Masking Description: Because interventions for the intervention group will be administered by the researcher, and participants will be aware that they are in the experimental group, blinding of researcher and participant is not possible. Statistical blinding will be ensured because coded data in the study will be analyzed by an independent statistician. Furthermore, blinding will be applied throughout the data collection and reporting processes to control reporting biases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group where simulation-supported training applications were performed (Experimental): Mothers will receive a six-week nursing intervention. The intervention will consist of four weeks of theoretical online training followed by two weeks of practical simulation training. The theoretical training will be planned according to Kolb's Experiential Learning Model and will be conducted in two sessions per week, with groups of 12 mothers per session. Additional sessions will be scheduled within the same week for mothers unable to attend.
  The theoretical training will cover topics such as first aid guidelines, preventing home accidents, parental supervision and first aid, identifying safety risks through image analysis, and watching relevant videos. Following the theoretical sessions, mothers will participate in four simulation scenarios over a two-week period. Each simulation will consist of a preliminary briefing, a simulation practice, and a debriefing session.
  Interventions: Other: Simulation based home accidents and first aid training program
- Control group that did not receive any training or simulation activity (No Intervention): The control group will not receive any intervention; mothers in this group will be measured three times: pretest, posttest, and follow up after three months. After the intervention group completes the interventions, the guidebook and videos will be shared with the control group.

INTERVENTIONS:
Other: Simulation based home accidents and first aid training program — The intervention is a six week nursing program designed to improve mothers knowledge and skills in preventing and managing home accidents.
  The intervention consists of researcher-supervised educational sessions, activities, and simulation based practices.
  Arms: The group where simulation-supported training applications were performed

SUMMARY:
Objective: This study will evaluate the effects of simulation-based nursing interventions on mothers of 2-4 year old children's ability to take safety precautions against home accidents, maintain parental supervision, and improve first aid knowledge and skills in home accidents.

Materials and Methods: This randomized, controlled experimental study will be conducted in accordance with the CONSORT 2025 guideline. A total of 48 mothers 24 in the intervention group and 24 in the control group residing in the Karatay district of Konya province and meeting the inclusion criteria will be included in the study. Data will be collected using an "Introductory Information Form," the "Safety Precautions for Children Aged 0-6 Scale," the "Parents' Supervisory Behavior Profile Scale," and the "First Aid Self Efficacy Scale for Home Accidents." Mothers in the intervention group will receive a six week nursing intervention consisting of a guidebook, educational sessions, video presentations, image analysis, and simulations. The control group will not receive any interventions. Post intervention, educational materials will be shared with the control group. Research data will be analyzed using SPSS 29 statistical software. Parametric and nonparametric tests based on normal distribution, analysis of variance, effect size, confidence interval, and Intention to Treat analyzes will be used for between group and within time comparisons.

Conclusion: The results of this study are expected to contribute to the development of evidence based educational practices to prevent home accidents, increase control skills, and strengthen first aid self efficacy in mothers.

ELIGIBILITY:
Inclusion Criteria:

* Mother with at least primary school education
* Having a healthy child aged 2-4 years
* Volunteering to participate

Exclusion Criteria:

* Child's previous hospitalization due to a home accident
* Home accident/first aid training in the last year
* Maternal psychiatric diagnosis
* Mother being employed
* Child in poor health Mother being an immigrant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers
Enrollment: 48 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Scale for diagnosing mothers safety precautions against home accidents in children aged 0-6 | 6 weeks
  The scale was developed to determine the safety precautions taken by mothers of children aged 0-6 to protect their children from home accidents. The 5-point Likert-type scale consists of 40 items, 34 positive and 6 negative (items 6, 9, 23, 26, 30, and 40). Positive items are scored as Always (5), Most of the Time (4), Sometimes (3), Rarely (2), and Never (1); and negative items are scored as Always (1), Most of the Time (2), Sometimes (3), Rarely (4), and Never (5). The highest possible score is 200, and the lowest is 40. Higher scores indicate that mothers take the highest level of precautions to protect themselves from home accidents. Cronbach's alpha for the study is 0.82.
Parents Supervisory Behavior Profile Scale | 6 weeks
  The scale aims to measure the risk of unintentional injury to children aged 2-5 under parental supervision. The scale has a 5-point Likert-type structure. Each item is scored from 1 to 5. Negatively worded items (items 13 and 17) are reverse-coded. The scale consists of 29 items and four subscales: protectiveness (9 items), supervision needs (9 items), risk tolerance (8 items), and belief that fate controls the child's health (3 items). The internal consistency coefficient of the scale is 0.75, and the subscales range from 0.57 to 0.79.
First Aid Self Efficacy Scale for Home Accidents | 6 weeks
  The scale determines the first aid self-efficacy levels of mothers of children aged 0-4 in the event of a home accident. The scale consists of 12 items with a 5-point Likert-type structure and a single dimension. Responses are scored as follows: Strongly agree (5), Agree (4), Undecided (3), Disagree (2), and Strongly disagree (1). The highest possible score is 60; the lowest is 12. Higher scores indicate increased self-efficacy in first aid. The study's Cronbach's alpha was 0.84.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Selçuklu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Personally, I don't prefer this situation.

REFERENCES:
- [Background] Wei YL, Chen LL, Li TC, Ma WF, Peng NH, Huang LC. Self-efficacy of first aid for home accidents among parents with 0- to 4-year-old children at a metropolitan community health center in Taiwan. Accid Anal Prev. 2013 Mar;52:182-7. doi: 10.1016/j.aap.2012.12.002. Epub 2013 Jan 21. PMID 23348100
- [Background] Gallagher L, Breslin G, Leavey G, Curran E, Rosato M. Determinants of unintentional injuries in preschool age children in high-income countries: A systematic review. Child Care Health Dev. 2024 Jan;50(1):e13161. doi: 10.1111/cch.13161. Epub 2023 Aug 9. PMID 37555597
- [Background] Bai P, Zang X, Liu R, Wang L, Dai C, Yang G. In-situ simulation for nursing students' professional competence development in postanesthesia care: A quasi-experimental study. Nurse Educ Pract. 2023 Jul;70:103660. doi: 10.1016/j.nepr.2023.103660. Epub 2023 May 9. PMID 37178479
- [Background] Jullien S. Prevention of unintentional injuries in children under five years. BMC Pediatr. 2021 Sep 8;21(Suppl 1):311. doi: 10.1186/s12887-021-02517-2. PMID 34496772